CLINICAL TRIAL: NCT04860336
Title: Glycemic Observation and Metabolic Outcomes in Mothers and Offspring / Glycemic Profile of Pregnancy Consortium
Brief Title: Glycemic Observation and Metabolic Outcomes in Mothers and Offspring
Acronym: GO MOMs
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Yale University (Other); Women and Infants Hospital of Rhode Island (Other); University of Pittsburgh (Other); Massachusetts General Hospital (Other); Tufts Medical Center (Other); Columbia University (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Denise Scholtens, Professor, Northwestern University
Other Study IDs: GO MOMs; 1U01DK123759-01 (NIH); 5U01DK123759-02 (NIH); 3U01DK123759-01S1 (NIH); 1U01DK123783-01 (NIH); 1U01DK123791-01 (NIH); 1U01DK123795-01 (NIH); 1U01DK123745-01 (NIH); 1U01DK123799-01 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes; Pregnancy Related
Keywords: gestational diabetes; continuous glucose monitor; oral glucose tolerance test; gestational diabetes mellitus; GDM; OGTT; CGM; glucose tolerance test; glycemic regulation; pregnancy; large for gestational age; observational
MeSH Terms: conditions — Diabetes, Gestational | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants are given the option to have blood collected for future DNA analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pregnant women less than or equal to 14w0d gestation
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The overarching goal of Glycemic Observation and Metabolic Outcomes in Mothers and Offspring (GO MOMs) is to perform a comprehensive, longitudinal description of maternal glycemia over the course of pregnancy and to evaluate how glucose levels throughout pregnancy relate to traditional third trimester gestational diabetes mellitus (GDM) screening and perinatal outcomes.

DETAILED DESCRIPTION:
GO MOMs is an observational study designed to characterize the glycemic profile of pregnancy using continuous glucose monitoring (CGM) technology in order to develop criteria using CGM measurements and/or early pregnancy oral glucose tolerance testing (OGTT) at 10w0d-14w0d gestation that are predictive, along with clinical factors, of adverse pregnancy outcomes in mothers and their newborns. GO MOMs involves multiple institutions and an anticipated 2179 participants. Participants will attend 4 research study visits: Visit 1 (10w0d-14w0d gestation), Visit 2 (16w0d-20w0d gestation), Visit 3 (24w0d-28w0d gestation), and Visit 4 (32w0d-36w0d gestation). Additional data will be collected at a Delivery Visit and via chart abstraction. Mothers will have a Remote Follow-up call after delivery to collect additional data. At Visits 1-4, a blinded CGM sensor will be placed. Participants will be instructed to wear the sensor for 10 days after which time they will follow instructions to return it to their study site. At Visit 1 (10w0d-14w0d gestation), participants will undergo a 75 g 2-hour (hr) OGTT. At Visit 3 (24w0d-28w0d gestation), participants will undergo a 100 g 3 hr OGTT. Visit 1 will include an extended maternal interview to collect social and demographic, medical history, obstetrical history, surgical history, family medical history, current health and pregnancy, and lifestyle (sleep, alcohol, tobacco use) data. Medical history, alcohol and tobacco use data will be updated at each study visit. Sleep data will be updated at Visit 3 (24w0d-28w0d gestation). Blood and urine samples will also be obtained at each visit for additional laboratory testing and some will be stored for ancillary investigations. At the Delivery Visit, newborn physical measurements including weight, length and skinfolds will be performed. Birthweight at delivery will also be obtained through chart abstraction. Primary statistical analyses will be performed to develop predictive criteria based on CGM and/or OGTT measures at Visit 1 (10w0d-14w0d gestation) along with clinical factors for primary maternal and newborn outcomes. Secondary analyses will further refine predictive models and will evaluate associations of maternal glucose with secondary outcomes and longitudinal modeling of maternal glycemia over the course of pregnancy.

GO MOMs Nutrition Substudy: The GO MOMs Nutrition Study is an observational substudy nested within the GO MOMs parent study. The goal of the study is to describe self-reported dietary components in a diverse cohort of pregnant individuals and to study the relationship between maternal diet and outcomes including maternal glycemia, maternal insulin physiology, infant birth weight, and infant fat mass. Participants will complete 6 dietary recalls via the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool during their pregnancies (Figure). Two will occur at visits and four will be unannounced, meaning they are completed on a random day without advance notice, during CGM wear. In addition, stored samples from all GO MOMs participants at visit 1 and 3 will be assayed for other nutritional markers. Primary statistical analyses will be used to identify associations between dietary carbohydrate content at <22 weeks' gestation and maternal glycemia 24-28 weeks' gestation and neonatal birthweight.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age >=18 at consent
* Singleton gestation
* 10w0d-14w0d gestation at the time of the Visit 1 OGTT and CGM placement according to study dating criteria
* Conceived using own oocyte
* Willing and able to wear CGM as directed and adhere to CGM instructions
* Planning to deliver at GO MOMs-affiliated hospital (see list of accrual sites in the protocol section "Key Roles and Contact Information").

Exclusion Criteria:

* Pre-existing diabetes at enrollment
* Currently self-monitoring blood glucose
* Current use of medication with glycemic effects
* Fetal malformation evident at or before enrollment that is likely lethal. This includes, but is not limited to, malformations such as anencephaly, hydrops, diffuse subcutaneous edema or cystic hygroma, ectopic cordis, and encephalocele
* Known fetal aneuploidy based on chorionic villus sampling
* Participation in other research study that may modify glycemic profile or study outcomes
* History of bariatric surgery
* Extensive skin changes or diseases making CGM sensor use problematic
* Significant allergy to adhesive
* Previous participation in GO MOMs
* Current bulimia or anorexia nervosa
* Overnight shift work that alters the sleep/wake periods
* Hemoglobin A1c >= 6.5%, fasting glucose >= 126 mg/dL or 2 hr glucose >= 200 mg/dL noted during OGTT at 10w0d-14w0d gestation
* Current psychiatric illness/social situation that would limit compliance with study requirements, as determined by the site investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant adults who enroll prior to 10w0d-14w0d gestation.
Sampling Method: Non-Probability Sample
Enrollment: 2179 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes (GDM) | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Primary outcome in GO MOMs mothers: Number of mothers diagnosed with gestational diabetes mellitus (GDM) using a 100 g 3 hr OGTT at 24w0d-28w0d gestation according to Carpenter-Coustan criteria (at least two of the timed glucose measurements greater than or equal to the following thresholds: fasting >= 95 mg/dL, 1 hr >= 180 mg/dL, 2 hr >= 155 mg/dL, 3 hr >= 140 mg/dL).
Large for gestational age (LGA) | Delivery
  Primary outcome in GO MOMs newborns: Number of newborns who are large for gestational age (LGA), defined as birthweight >90th percentile for gestational age according to Aris et al. (2019). The first birthweight after delivery obtained from medical chart abstraction will be used for defining the primary LGA outcome.

SECONDARY OUTCOMES:
Hypertension | Evaluated 30-90 days after delivery through chart abstraction for any events occurring during pregnancy
  Secondary outcome in GO MOMs mothers: Number of mothers with hypertensive disorders of pregnancy including preeclampsia with and without severe features, gestational hypertension, eclampsia, and Hemolysis, Elevated Liver enzymes, and Low Platelet count (HELLP) syndrome, defined by the American College of Obstetricians and Gynecologists (ACOG) criteria
Cesarean delivery | Delivery
  Secondary outcome in GO MOMs mothers: Number of mothers with cesarean delivery
Sum of skinfolds | Within 72 hours after delivery
  Secondary outcome in GO MOMs newborns: Newborn sum of flank, triceps, and subscapular skinfolds, evaluated as a continuous measure and dichotomized as >90th percentile.
Small for gestational age (SGA) | Delivery
  Secondary outcome in GO MOMs newborns: Number of newborns who are small for gestational age (SGA), defined as birthweight < 10th percentile for gestational age according to Aris et al. (2019)
Preterm birth | Delivery
  Secondary outcome in GO MOMs newborns: Number of newborns with preterm birth, defined as delivery prior to estimated gestational age 37 weeks 0 days.
Shoulder dystocia | Delivery
  Secondary outcome in GO MOMs newborns: Number of newborns with shoulder dystocia, identified through chart abstraction and defined clinically, requiring documentation that providers applied maneuvers to reduce the shoulder at delivery.
Neonatal birth injury | Delivery
  Secondary outcome in GO MOMs newborns: Number of newborns with neonatal birth injury, identified through chart abstraction and defined as brachial plexus palsy or clavicular, humeral, or skull fracture.
Neonatal hypoglycemia | Within 30 days after delivery
  Secondary outcome in GO MOMs newborns: Number of newborns with neonatal hypoglycemia, identified through chart abstraction and defined as treated neonatal hypoglycemia.
Neonatal respiratory morbidity | Within 30 days after delivery
  Secondary outcome in GO MOMs newborns: Number of newborns with neonatal respiratory morbidity, identified through chart abstraction and defined as need for respiratory support within 72 hrs after birth and consisting of one or more of the following: the use of continuous positive airway pressure (CPAP) or high-flow nasal cannula for at least 2 consecutive hrs, supplemental oxygen with a fraction of inspired oxygen of at least 0.30 for at least 4 continuous hrs, extracorporeal membrane oxygenation (ECMO), or mechanical ventilation. A high flow of air or blended air and oxygen is defined as more than 1 liter per minute
Neonatal hyperbilirubinemia | Within 30 days after delivery
  Secondary outcome in GO MOMs newborns: Number of newborns with neonatal hyperbilirubinemia, identified through chart abstraction and defined as treatment of hyperbilirubinemia in the first week of life with phototherapy or exchange transfusion or a diagnosis of kernicterus.
Nutrition Substudy: Mean CGM glucose in mothers | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Outcome in mothers for Nutrition Substudy: Mean CGM glucose at 24-28 weeks' gestation in mothers
Nutrition Substudy: Percent time above various glycemic thresholds at 24-28 weeks | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Secondary outcome in mothers for Nutrition Substudy: Percent time above various glycemic thresholds: 100 miligrams/deciliter, 105 miligrams/deciliter, 110 miligrams/deciliter, 120 miligrams/deciliter, 140 miligrams/deciliter, as measured by continuous glucose monitor at 24-28 weeks' gestation.
Nutrition Substudy: Mean nocturnal glucose | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Secondary outcome in mothers for Nutrition Substudy: Mean nocturnal glucose (12am-6am) in miligrams/deciliter, as measured by continuous glucose monitor at 24-28 weeks' gestation.
Nutrition Substudy: Percent time above various glycemic thresholds at 16-36 weeks | When participants are between 16 weeks 0 days pregnant to 36 weeks 0 days pregnant
  Secondary outcome in mothers for Nutrition Substudy: Maternal continuous glucose monitor-assessed glucose defined as percent time above various glycemic thresholds: 100 miligrams/deciliter, 105 miligrams/deciliter, 110 miligrams/deciliter, 120 miligrams/deciliter, 140 miligrams/deciliter, as measured by continuous glucose monitor at 16-20, 24-28, and 32-36 weeks' gestation.
Nutrition Substudy: Insulin resistance | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Secondary outcome in mothers for Nutrition Substudy: Insulin resistance, as estimated by the Matsuda index quantified during the oral glucose tolerance test at 24-28 weeks' gestation. The Matsuda index calculates whole body insulin resistance, with insulin resistance defined as being equal to or lower than 2.5.
Nutrition Substudy: Insulin secretory response | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Secondary outcome in mothers for Nutrition Substudy: Insulin secretory response, as estimated by the ratio of insulin area under the curve to glucose area under the curve, during oral glucose tolerance test at 24-28 weeks' gestation.
Nutrition Substudy: gestational diabetes mellitus diagnosis | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Secondary outcome in mothers for Nutrition Substudy: Gestational diabetes mellitus, diagnosed using Carpenter-Coustan criteria applied to an oral glucose tolerance test at 24-28 weeks' gestation.
Nutrition Substudy: Neonatal fat mass | Within 72 hours of delivery
  Secondary outcome in newborns for Nutrition Substudy: Neonatal fat mass as estimated by flank skinfold, measured as percent body fat, within 72 hours of delivery.
Nutrition Substudy: large for gestational age birthweight | Delivery
  Secondary outcome in newborns for Nutrition Substudy: Large for gestational age birth weight defined as birth weight > 90th percentile for gestational age.
Nutrition Substudy: Birthweight for gestational age percentile | Delivery
  Secondary outcome for newborns for Nutrition Substudy: Birthweight for gestational age percentile. The first weight after delivery from the medical record will be used for defining this outcome.

OTHER OUTCOMES:
Neonatal intensive care unit (NICU) admissions | Within 30 days after delivery
  Exploratory outcome in GO MOMs newborns: Number of newborns with neonatal intensive care unit (NICU) admissions
Length of hospital admission | Within 30 days after delivery
  Exploratory outcome in GO MOMs newborns: Length of admission/length of stay (for NICU or entire delivery hospitalization) for newborns
Spontaneous abortion | Prior to 20 weeks' gestation
  Exploratory outcome in GO MOMs mothers: Spontaneous abortion (< 20 weeks of gestation)
Stillbirth | Delivery
  Exploratory outcome in GO MOMs newborns: Number of mothers with stillbirth (intrauterine fetal demise at 20 weeks of gestation or later)
Neonatal death | Within 30 days after delivery
  Exploratory outcome in GO MOMs newborns: Number of newborns with neonatal death
Major congenital malformation | Within 30 days after delivery
  Exploratory outcome in GO MOMs newborns: Number of newborns with major congenital malformation
Antepartum admissions or maternal readmissions | Within 30 days after delivery
  Exploratory outcome in GO MOMs mothers: Number of mothers with antepartum admissions or maternal readmissions
Apgar score <7 at 5 minutes | Delivery
  Exploratory outcome in GO MOMs newborns: Number of newborns with Apgar score <7 at 5 minutes
Nutrition Substudy: Maternal fasting triglycerides | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Exploratory outcome in mothers for Nutrition Substudy: Maternal fasting triglycerides as measured in miligrams/deciliter at 24-28 weeks' gestation.
Nutrition Substudy: Maternal fasting free fatty acids | When participants are between 24 weeks 0 days pregnant to 28 weeks 0 days pregnant
  Exploratory outcome in mothers for Nutrition Substudy: Maternal fasting free fatty acids as measured in millimoles per liter at 24-28 weeks' gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Scholtens, PhD, Principal Investigator — Northwestern University
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Kaiser Permanente - Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - Kaiser Permanente - Northwest, Portland, Oregon
  - Magee Womens Research Institute & Foundation, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Participants have the option to agree to share dataset with National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Repository.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] GO MOMs Study Group. Design, rationale and protocol for Glycemic Observation and Metabolic Outcomes in Mothers and Offspring (GO MOMs): an observational cohort study. BMJ Open. 2024 Jun 8;14(6):e084216. doi: 10.1136/bmjopen-2024-084216. PMID 38851233
- See also: Information about the study — http://www.gomomsstudy.org